CLINICAL TRIAL: NCT03147547
Title: Participation in Preventive Parenting Interventions
Brief Title: Parent Engagement Package: Initial Testing of Strategies to Increase Participation in Parenting Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: J.B. Sutton Elementary School (Unknown)
Responsible Party: Principal Investigator, Emily Winslow PhD, Assistant Research Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0812003515
Record Dates: First submitted 2017-04-18; First posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Patient Compliance
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two conditions: 1) promotional brochure plus an attention-control research interview or 2) Package Engagement Package
Who Masked: Participant
Masking Description: single-blind masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Promotional Brochure (Active Comparator): Participants in this condition received one of the strategies in the Parent Engagement Package: a promotional brochure with information about the parenting intervention being offered at their child's school, the Triple P Positive Parenting Program. This information included the location of meetings, free childcare, topics covered, choice of English or Spanish groups, meeting day and time, and an enrollment form. Parents who returned the enrollment form received a confirmation letter prior to the first parenting program session.
  Interventions: Other: Promotional Brochure
- Parent Engagement Package (Experimental): Participants in this condition received all engagement strategies in the Parent Engagement Package, which included: 1) the promotional brochure; 2) family testimonial flyer that included photos and quotes from prior participants; 3) teacher endorsement of the Triple P program; 4) provider engagement call to motivate parents to attend; and 5) phone reminders prior to each Triple P session.
  Interventions: Other: Promotional Brochure; Other: Family Testimonial Flyer; Other: Teacher Endorsement; Other: Provider Engagement Call

INTERVENTIONS:
Other: Promotional Brochure — Promotional brochure with information about the Triple P Positive Parenting Program and an enrollment form.
Other: Family Testimonial Flyer — Flyer that included quotes and photos from parents who had previously participated in the Triple P Positive Parenting Program and/or their children who participated in the free childcare.
  Arms: Parent Engagement Package
Other: Teacher Endorsement — Brief conversation between the parent and their child's teacher in which the teacher told the parent about the benefits of participating in the Triple P Positive Parenting Program and recommended the parent attend.
  Arms: Parent Engagement Package
Other: Provider Engagement Call — This was a manualized, 20-minute call from the Triple P Positive Parenting Program provider to a parent in which the provider elicited the parent's child-focused goals and showed how the parent's goals could be addressed by Triple P. The provider also helped the parent problem solve barriers to attendance and develop an action plan to handle common barriers (e.g., scheduling conflicts) as well as set session reminders.
  Arms: Parent Engagement Package

SUMMARY:
This study evaluated the effectiveness of strategies for engaging parents into parenting programs. Engagement strategies included a booklet showing testimonial quotes and photos from prior participants, a recommendation to attend for the child's teacher, and a motivational call from the parenting program provider. It was hypothesized that the combination of engagement strategies would increase attendance at a parenting intervention compared to receiving only a promotional brochure and research interview.

ELIGIBILITY:
Inclusion Criteria:

* Is the biological or adoptive mother of a child in kindergarten or 3rd grade at the participating school (i.e., "target child");
* The target child lived with the mother at least half of the time;
* The mother spoke English or Spanish;

Exclusion Criteria:

* The target child changed schools;
* The mother reported the target child would be changing schools during the school year;
* The target child attended one of the participating schools during a previous cohort of the study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — To be eligible, a caregiver had to self-report that she was the biological or adoptive mother of the target child (i.e., the child in kindergarten or 3rd grade at the participating school).
Enrollment: 122 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Parenting Intervention Attendance | Attendance was recorded by Triple P providers at each session, once per week for 8 weeks
  Number of sessions a caregiver from a student's family attended the parenting intervention, the Triple P Positive Parenting Program

SECONDARY OUTCOMES:
Parenting Intervention Enrollment | from the date engagement strategies commenced until the date the Triple P Positive Parenting Program began, up to 7 weeks
  Whether or not a family enrolled in the Triple P Positive Parenting Program by completing an enrollment form or answering 'yes' to an enrollment question during the provider engagement call or attention-control research interview
Parenting Intervention Homework Completion | collected once per week for 7 weeks, at the beginning of each Triple P Positive Parenting Program sessions 2 through 8
  Caregiver report of completion of Triple P Positive Parenting Program assignments between sessions
Parenting Intervention Session Involvement | collected once per week for 8 weeks, after each Triple P Positive Parenting Program session
  Provider reports of the extent to which a caregiver actively participated in each Triple P Positive Parenting Program session attended
Child Behavior Problems | collected 1 week before Triple P session 1 and at Triple P post-test, which was 9 weeks after the first behavior reports were collected
  Teacher report of child behavior in the classroom

CONTACTS AND LOCATIONS:
Overall Officials: Emily B Winslow, Ph.D., Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Winslow EB, Poloskov E, Begay R, Tein JY, Sandler I, Wolchik S. A randomized trial of methods to engage Mexican American parents into a school-based parenting intervention. J Consult Clin Psychol. 2016 Dec;84(12):1094-1107. doi: 10.1037/ccp0000140. Epub 2016 Sep 5. PMID 27599226